CLINICAL TRIAL: NCT04583579
Title: Maximizing the Initial Experience of a Neophyte Scleral Lens Wearer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator ended full-time appointment at university.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Pucker, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300006015
Record Dates: First submitted 2020-09-23; First posted 2020-10-12 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Contact Lens Adaptation
Keywords: Contact Lenses; Scleral Lenses; Adaptation; Neophyte

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to try all five scleral lens application methods in a random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- New Scleral Lens Wearers (Experimental): All patients will be asked to wear scleral lenses for the duration of this study.
  Interventions: Device: DMV inserter (DMV® MagicTouch™) with an open end; Device: DMV inserter (DMV® MagicTouch™) with a closed end; Device: Three fingers (Patient's Hand); Device: O-ring (Hardware Store Product); Device: Tea light candle (Generic Deparment Store Product) with DMV inserter (DMV® MagicTouch™)

INTERVENTIONS:
Device: DMV inserter (DMV® MagicTouch™) with an open end — This is a device used to help apply scleral lenses.
Device: DMV inserter (DMV® MagicTouch™) with a closed end — This is a device used to help apply scleral lenses.
Device: Three fingers (Patient's Hand) — This is a device used to help apply scleral lenses.
Device: O-ring (Hardware Store Product) — This is a device used to help apply scleral lenses.
Device: Tea light candle (Generic Deparment Store Product) with DMV inserter (DMV® MagicTouch™) — This is a device used to help apply scleral lenses.

SUMMARY:
The goal of this proposal is to conduct a randomized controlled study aimed at learning the best method for applying scleral lenses and factors associated with successfully completing scleral lens application and removal training.

DETAILED DESCRIPTION:
Scleral lens (SL) prescribing has dramatically increased over the past few years likely because of the advent of better SL designs, better materials, and greater awareness of the technology. SL market growth has also likely increased because SLs were once reserved for patients with complex ocular surface diseases, though advances with SL technologies have allowed SL fitting to include patients with dry eye and even patients who have relatively uncomplicated refractive errors. While SLs are maintained and cared for much like soft contact lenses (e.g., they require a contact lens care system), SL wearers also need help with applying their lenses. Patients specifically are advised by their care provider to insert their SLs with their fingers (tripod method), a DMV inserter with an open or closed end (hole potentially aides in vision), or a specialized o-ring that is balanced on a finger. Our clinic also utilizes a tea light candle with a DMV inserter attached to the top of it when patients have mobility issues. While work from this investigator's study group has found that 54% of patients prefer DMV inserters for applying their SLs as compared to the above other options, these preliminary data were obtained through a cross-sectional electronic survey from subjects who completed their SL fitting up to two years ago. Therefore, the goal of this proposal is to conduct a randomized controlled study aimed at learning the best method for applying SLs and factors associated with successfully completing SL application and removal training. These data are needed because it will help practitioners with patient education and because it may increase the likelihood that patients will be successful with SLs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Must have an indication for needing scleral lenses

Exclusion Criteria:

* Participating in another research study
* Unable to attend multiple visits
* Advanced knowledge or past use of scleral lenses
* A physical or mental condition that would prevent the subject from applying their own scleral lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to sure individual participant data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Scleral Lens Wearers
Started | 17
Completed | 13
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | New Scleral Lens Wearers
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (20.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Scleral Lens Application Time
Description: Amount of time needed to apply scleral lenses to both eyes (minutes); each patient will try each application method in a random order.
Time Frame: At Dispense Visit at Hour 0 (Visit 2)
Population: Each subject tried all 5 methods.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With an Open End: DMV inserter (DMV® MagicTouch™) with an open end: This is a device used to help apply scleral lenses.
- New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With a Closed End: DMV inserter (DMV® MagicTouch™) with a closed end: This is a device used to help apply scleral lenses.
- New Scleral Lens Wearers - Three Fingers (Patient's Hand): Three fingers (Patient's Hand): This is a device used to help apply scleral lenses.
- New Scleral Lens Wearers - O-ring (Hardware Store Product): O-ring (Hardware Store Product): This is a device used to help apply scleral lenses.
- New Scleral Lens Wearer - Tea Light Candle (Generic Deparment Store Product) With DMV Inserter: Tea light candle (Generic Deparment Store Product) with DMV inserter (DMV® MagicTouch™): This is a device used to help apply scleral lenses.
Arm/Group | New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With an Open End | New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With a Closed End | New Scleral Lens Wearers - Three Fingers (Patient's Hand) | New Scleral Lens Wearers - O-ring (Hardware Store Product) | New Scleral Lens Wearer - Tea Light Candle (Generic Deparment Store Product) With DMV Inserter
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
minutes | 75.2 (20.7) | 71.6 (25.9) | 51.3 (38.5) | 62.5 (37.5) | 63.9 (35.7)
Statistical Analysis 1: Comparison: New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With an Open End vs New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With a Closed End vs New Scleral Lens Wearers - Three Fingers (Patient's Hand) vs New Scleral Lens Wearers - O-ring (Hardware Store Product) vs New Scleral Lens Wearer - Tea Light Candle (Generic Deparment Store Product) With DMV Inserter; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Subject's Method Preference
Description: Patient top ranked preference of scleral lens application method (percent)
Time Frame: At Dispense Visit at Hour 0 (Visit 2)
Measure: Count of Participants; unit: Participants
Arm/Group | New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With an Open End | New Scleral Lens Wearers - DMV Inserter (DMV® MagicTouch™) With a Closed End | New Scleral Lens Wearers - Three Fingers (Patient's Hand) | New Scleral Lens Wearers - O-ring (Hardware Store Product) | New Scleral Lens Wearer - Tea Light Candle (Generic Deparment Store Product) With DMV Inserter
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
Participants | 1 | 5 | 1 | 2 | 4

ADVERSE EVENTS:
Time Frame: About 3 months
Groups:
- New Scleral Lens Wearers: All subjects will be asked to wear scleral lenses for the duration of this study. All subjects tried all interventions during the same session, so it is not possible to separate subjects into different groups. Each subject tried the following interventions on the same day within minutes of each other:
  DMV inserter (DMV® MagicTouch™) with an open end: This is a device used to help apply scleral lenses.
  DMV inserter (DMV® MagicTouch™) with a closed end: This is a device used to help apply scleral lenses.
  Three fingers (Patient's Hand): This is a device used to help apply scleral lenses.
  O-ring (Hardware Store Product): This is a device used to help apply scleral lenses.
  Tea light candle (Generic Deparment Store Product) with DMV inserter (DMV® MagicTouch™): This is a device used to help apply scleral lenses.
Arm/Group | New Scleral Lens Wearers
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04583579/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04583579/ICF_002.pdf